CLINICAL TRIAL: NCT06817356
Title: A Phase 2, Double-Blind, Proof of Concept Study to Evaluate Mazdutide Compared With Placebo in Participants With Alcohol Use Disorder
Brief Title: A Study to Evaluate Mazdutide Compared With Placebo in Participants With Alcohol Use Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 27290; I8P-MC-OXAH (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-02-05; First posted 2025-02-10 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — mazdutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mazdutide (Experimental): Mazdutide administered subcutaneously (SC).
  Interventions: Drug: Mazdutide
- Placebo (Placebo Comparator): Placebo administered SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mazdutide — Administered SC
  Other Names: LY3305677
  Arms: Mazdutide
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The objective of this proof-of-concept study to evaluate mazdutide in participants with alcohol use disorder (AUD).

For any individual participant, the maximum duration of study participation is approximately 36 weeks, including screening and posttreatment follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Current AUD diagnosis as defined by Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 criteria.

Exclusion Criteria:

* Have a history of significant active or unstable major depressive disorder, suicidal ideation, or other severe psychiatric disorder within the last 12 months.
* Have initiated psychotherapy, changed the intensity of psychotherapy, or other nondrug therapies (for example, acupuncture or hypnosis) within 8 weeks prior to enrollment.
* Have received any medication for AUD in the last 30 days including but not limited to, disulfiram, acamprosate, naltrexone, gabapentin, baclofen, or topiramate.
* Other protocol-specific inclusion and exclusion criteria may apply.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Behaviors Associated with Alcohol Use Disorder (AUD) as Assessed by the Timeline Followback Method | Baseline, Week 28

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (27):
- United States (27):
  - Headlands Research - Scottsdale, Scottsdale, Arizona
  - Woodland International Research Group, Little Rock, Arkansas
  - Woodland Resarch Northwest/ERG, Rogers, Arkansas
  - Ark Clinical Research - Fountain Valley, Fountain Valley, California
  - Synergy San Diego, Lemon Grove, California
  - Headlands Research-Artemis San Diego, San Diego, California
  - Research Centers of America ( Hollywood ), Hollywood, Florida
  - K2 Medical Research - Maitland, Maitland, Florida
  - K2 Medical Research, Maitland, Florida
  - Clinical Neuroscience Solutions Inc, Orlando, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - K2 Medical Research - Tampa, Tampa, Florida
  - CenExel iResearch, LLC (CenExel iRA), Decatur, Georgia
  - DelRicht Research, Mandeville, Louisiana
  - Adams Clinical, Watertown, Massachusetts
  - Vitalix Clinical, Worcester, Massachusetts
  - Redbird Research LLC, Las Vegas, Nevada
  - IMA Clinical Research Albuquerque, Albuquerque, New Mexico
  - Richmond Behavioral Associates, Staten Island, New York
  - Ichor Research, Syracuse, New York
  - Davis Clinical, The Bronx, New York
  - Summit Headlands, Portland, Oregon
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Clinical Neuroscience Solutions Inc, Memphis, Tennessee
  - FutureSearch Trials of Dallas, Dallas, Texas
  - Dallas Clinical Research Center/Pillar Research, Richardson, Texas

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/